CLINICAL TRIAL: NCT02366403
Title: Breathing Meditation Intervention for Post-Traumatic Stress Disorder
Brief Title: Breathing Meditation Intervention for Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1485-R; IRX001485A (Other Grant/Funding Number: Dept. of Veterans Affairs)
Record Dates: First submitted 2015-01-12; First posted 2015-02-19 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Meditation; Yoga; Cognitive Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SKY (Experimental): a standardized meditation program
  Interventions: Behavioral: SKY meditation
- CPT-C (Active Comparator): CPT-C (Cognitive Processing Therapy-cognitive only) is a standardized, manual-based treatment consisting of 12, 60-minute sessions which will be given twice per week. Sessions will focusing on specific issues, learning new therapeutic techniques and setting up homework for the following session including real-life application of learned CPT techniques.
  Interventions: Behavioral: CPT-C

INTERVENTIONS:
Behavioral: SKY meditation — SKY (Sudarshan Kriya Yoga) meditation is a standardized, manual-based and replicable program that includes relaxation techniques as well as periods of discussion. The format is a 7-day intensive group class (2 1/2 hours/day intensive format) followed by five weeks of sessions twice per week (1hr/session). SKY meditation incorporates several types of breathing exercises involving arousal and attentional control. Initial breathing exercises are calming and focusing. Subsequent breathing exercises are more fully engaging energizing, allowing the practitioner to focus more fully in each moment.
  Arms: SKY
Behavioral: CPT-C — CPT-C (Cognitive Processing Therapy-cognitive only) is a standardized, manual-based treatment consisting of 12, 60-minute sessions which will be given twice per week. Sessions will focusing on specific issues, learning new therapeutic techniques and setting up homework for the following session including real-life application of learned CPT techniques.
  Other Names: Cognitive Processing Therapy
  Arms: CPT-C

SUMMARY:
Post traumatic stress disorder (PTSD) is a condition that develops as a result of exposure to a traumatic event. The purpose of this study is to determine whether a breathing meditation technique (Sudarshan Kriya Yoga; SKY) provides a treatment benefit that is as effective as the standard intervention. Patients' PTSD symptoms will be monitored before treatment, at the end of treatment, one month after treatment and 12 months after treatment.

DETAILED DESCRIPTION:
Post traumatic stress disorder (PTSD) is a condition that develops as a result of exposure to a traumatic event and is characterized by intense physiological and psychological reactivity to stimuli associated with that trauma. PTSD represents a substantial proportion of the burden of illness among Veterans. A recent study found that PTSD was diagnosed in 13% of Veterans returning from Iraq and Afghanistan. Recent reports have also highlighted that PTSD is associated with suicidality - a fact that may explain the alarming rise of suicidal behavior amongst returning Veterans. Several studies suggest that meditation-based treatments may be helpful in treating PTSD. Sudarshan Kriya Yoga (SKY) is a meditation technique that involves a sequence of breathing exercises and has shown promise in treating PTSD. There are several lines of evidence to suggest that such meditation techniques provide a solid foundation for treating PTSD. First, breathing meditation techniques offer a powerful method for balancing autonomic nervous system activity that is often heightened in PTSD. Second, they promote the relaxation response that counters hyperarousal and results in a calmer approach to difficulties and challenges. Third, they may improve sleep quality. This may be important in treating PTSD because memories are encoded into long-term storage during sleep via a process known as consolidation. It is possible that the disturbed sleep which is common in PTSD (nightmares and insomnia) lead to disrupted memory consolidation. Therefore improvement in sleep may lead to improvement in PTSD.

Despite promising findings, meditation has not been sufficiently studied in Veterans to recommend its widespread use in treating PTSD. The goal of this proposal is to examine the effects of SKY meditation therapy on Veterans with clinically significant PTSD symptoms. SKY intervention will be compared to cognitive processing therapy (CPT) that is commonly used to treat Veterans with PTSD. CPT will be given as a "cognitive only" version (CPT-C) which is efficacious in treating PTSD. Veterans will be randomly assigned to one of the two groups (SKY, CPT-C; n=38 per group) and treatment will be delivered over a six-week period. A "noninferiority" experimental design will be used as is appropriate for trials in which the primary objective is to show that a novel intervention (SKY) is as effective as the standard intervention. Patients' PTSD symptoms will be monitored across time; before treatment (i.e., baseline), at the end of treatment, one month after treatment and 12 months after treatment. Other measures will be taken at baseline and at the end of treatment, and will include autonomic arousal (heart rate) and cognitive functioning including memory consolidation. The investigators will also monitor dropout rates as these can be high in conventional PTSD treatment programs. Based on preliminary studies using SKY in Veterans with PTSD and the existing literature, the investigators expect that PTSD symptom severity will be reduced following treatment with SKY, that this effect will not be clinically inferior to CPT-C and that the dropout rates will be no higher than CPT-C. Such findings would provide strong evidence for the efficacy of SKY in treating Veterans with PTSD. The investigators also expect that improvements in clinical measures of PTSD will correlate with improvements in memory consolidation, reflecting improvements in sleep following treatment. It is also likely that the individual's response to treatment will be influenced by their baseline characteristics. The SKY and CBT-C interventions focus on different aspects of PTSD; the SKY intervention focuses on breathing and relaxation techniques whereas CPT-C focuses on modifying the understanding of trauma through cognitive restructuring. For this reason the SKY intervention may be more effective for Veterans who have exaggerated arousal (e.g. heightened heart rate). In contrast the CPT-C intervention may be more effective for Veterans who have more cognitive symptoms (e.g., flashbacks, attentional difficulties) since CPT-C addresses cognitive processes. The long term goal of this project is to conduct a fully-powered multi-center randomized controlled clinical trial of SKY meditation in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veteran from any conflict era
* Symptoms of Posttraumatic Stress Disorder measured during study screening (scoring ≥38 on the PCL-5)

Exclusion Criteria:

* planning on starting a new course of behavioral therapy during the trial
* started new medication for PTSD within 8 weeks of the study screening
* participation in another study
* mania or psychosis within the past 6 months
* suicidal or homicidal intent within the past 60 days
* substance dependence (other than nicotine) within the past 30 days,
* seizure disorder
* severe traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Bayley, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 05/01/2020

REFERENCES:
- [Derived] Mathersul DC, Schulz-Heik RJ, Avery TJ, Allende S, Zeitzer JM, Bayley PJ. US Veterans Show Improvements in Subjective but Not Objective Sleep following Treatment for Posttraumatic Stress Disorder: Secondary Analyses from a Randomised Controlled Trial. Depress Anxiety. 2023 Aug 14;2023:7001667. doi: 10.1155/2023/7001667. eCollection 2023. PMID 40224604
- [Derived] Mathersul DC, Zeitzer JM, Schulz-Heik RJ, Avery TJ, Bayley PJ. Emotion regulation and heart rate variability may identify the optimal posttraumatic stress disorder treatment: analyses from a randomized controlled trial. Front Psychiatry. 2024 Feb 8;15:1331569. doi: 10.3389/fpsyt.2024.1331569. eCollection 2024. PMID 38389985
- [Derived] Bayley PJ, Schulz-Heik RJ, Tang JS, Mathersul DC, Avery T, Wong M, Zeitzer JM, Rosen CS, Burn AS, Hernandez B, Lazzeroni LC, Seppala EM. Randomised clinical non-inferiority trial of breathing-based meditation and cognitive processing therapy for symptoms of post-traumatic stress disorder in military veterans. BMJ Open. 2022 Aug 25;12(8):e056609. doi: 10.1136/bmjopen-2021-056609. PMID 36008059
- [Derived] Mathersul DC, Dixit K, Schulz-Heik RJ, Avery TJ, Zeitzer JM, Bayley PJ. Emotion dysregulation and heart rate variability improve in US veterans undergoing treatment for posttraumatic stress disorder: Secondary exploratory analyses from a randomised controlled trial. BMC Psychiatry. 2022 Apr 15;22(1):268. doi: 10.1186/s12888-022-03886-3. PMID 35428258
- [Derived] Mathersul DC, Tang JS, Schulz-Heik RJ, Avery TJ, Seppala EM, Bayley PJ. Study protocol for a non-inferiority randomised controlled trial of SKY breathing meditation versus cognitive processing therapy for PTSD among veterans. BMJ Open. 2019 Apr 3;9(4):e027150. doi: 10.1136/bmjopen-2018-027150. PMID 30948610

RESULTS

PARTICIPANT FLOW:
Groups:
- Sudarshan Kriya Yoga: a standardized meditation program
  SKY meditation: SKY (Sudarshan Kriya Yoga) meditation is a standardized, manual-based and replicable program that includes relaxation techniques as well as periods of discussion. The format is a 7-day intensive group class (2 1/2 hours/day intensive format) followed by five weeks of sessions twice per week (1hr/session). SKY meditation incorporates several types of breathing exercises involving arousal and attentional control. Initial breathing exercises are calming and focusing. Subsequent breathing exercises are more fully engaging energizing, allowing the practitioner to focus more fully in each moment.
Period: Overall Study
Arm/Group | Sudarshan Kriya Yoga | CPT-C
Started | 41 | 44
Completed | 30 | 29
Not Completed | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sudarshan Kriya Yoga | CPT-C | Total
Number analyzed (Participants) | 41 | 44 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (13.6) | 56.2 (11.7) | 56.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 34 | 41 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 31 | 57
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 23 | 29 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 41 | 44 | 85

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Checklist (PCL)
Description: Posttraumatic Stress Disorder Checklist-Civilian Version (PCL-C) (Blanchard et al., 1996) is a 17-item self- report scale that assesses PTSD symptom severity in the past month corresponding to DSM-IV criteria for PTSD. Scores range from 17-85 with higher scores reflecting greater severity. We used the civilian version to assess symptoms from both military and non-military trauma.
Time Frame: baseline, after treatment (six weeks), one month after treatment, and one year after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sudarshan Kriya Yoga | CPT-C
Number analyzed (Participants) | 41 | 44
score on a scale
  change from baseline to end of treatment | -5.6 (9.5) | -6.8 (11.4)
  change from baseline to one month after treatment | -4.8 (10.5) | -6.8 (11.9)
  change from baseline to one year after treatment | -4.4 (11.4) | -6.2 (10.7)

2. Secondary Outcome: Change in Beck Depression Inventory II (BDI-II)
Description: The BDI-II scale is a 21-item self-report measure that assesses depression symptom severity. Items are rated on a 4-point scale according to how much the symptom bothered the respondent over the prior two weeks. Scores range from 0-63 with higher scores reflecting greater severity.
Time Frame: baseline, after treatment (six weeks), one month after treatment, and one year after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sudarshan Kriya Yoga | CPT-C
Number analyzed (Participants) | 41 | 44
score on a scale
  Change from baseline to end of treatment | -6.1 (6.8) | -3.6 (10.9)
  Change from baseline to one month after treatment | -4.7 (8.7) | -2.8 (11.7)
  Change from baseline to one year after treatment | -5.6 (9.6) | -4.5 (10.0)

3. Secondary Outcome: Change in Positive and Negative Affect Schedule (PANAS)
Description: A 20-item self-report measure assessing positive and negative mood states over "the past few weeks" on a 5-point scale. Scores for positive and negative affect range from 10-50 with higher scores reflecting stronger affect.
Time Frame: baseline, after treatment (six weeks), one month after treatment, and one year after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sudarshan Kriya Yoga | CPT-C
Number analyzed (Participants) | 41 | 44
score on a scale
  PANAS positive: change from baseline to end of treatment | 2.5 (5.8) | 0.3 (5.9)
  PANAS positive: change from baseline to one month after treatment | 1.3 (8.6) | -1.3 (7.1)
  PANAS positive: change from baseline to one year after treatment | -0.1 (10.5) | 0.4 (7.0)
  PANAS negative: change from baseline to end of treatment | -3.2 (4.6) | -0.9 (8.8)
  PANAS negative: change from baseline to one month after treatment | -2.9 (6.7) | -1.2 (8.4)
  PANAS negative: change from baseline to one year after treatment | -1.8 (8.2) | -1.7 (8.0)

ADVERSE EVENTS:
Time Frame: baseline to one year posttreatment (i.e. 58 weeks)
Description: Study staff conducted safety evaluations and followed safety protocols whenever a participant endorsed any suicidal or homicidal ideation, including via self report measures.
Arm/Group | Sudarshan Kriya Yoga | CPT-C
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/44
Other Adverse Events (participants affected / at risk) | 0/41 | 1/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sudarshan Kriya Yoga (N=41) | CPT-C (N=44)
Admission to inpatient psychiatry (Psychiatric disorders) | 0 (0) | 1 (1) — One participant presented to the emergency room with suicidal ideation and was admitted to inpatient psychiatry.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sudarshan Kriya Yoga (N=41) | CPT-C (N=44)
Distressed and lost to follow up (Psychiatric disorders) | 0 (0) | 1 (1) — One participant reported being distressed by the written assignments and was lost to follow up. The study's safety protocol was followed and the participant was determined to not be at imminent risk of harm.

LIMITATIONS AND CAVEATS:
SKY involved more hours of instruction than CPT (25 vs 12 hours).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02366403/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT02366403/SAP_001.pdf